CLINICAL TRIAL: NCT00560573
Title: Phase 1, Dose Escalation Study Of CP-751,871 In Combination With Cisplatin And Gemcitabine In Previously Untreated Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Study Of CP-751,871 In Combination With Cisplatin And Gemcitabine In Chemotherapy-Naïve Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4021015
Record Dates: First submitted 2007-11-15; First posted 2007-11-19 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — figitumumab; Cisplatin; Gemcitabine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: CP-751,871; Drug: Cisplatin; Drug: Gemcitabine; Drug: Pemetrexed

INTERVENTIONS:
Drug: CP-751,871 — CP-751,871 at doses ranging from 6 to 20 mg/Kg on Day 1 of each 21-day cycle. CP-751,871 may be administered even after active comparators discontinuation, for a total number of 17 cycles (1 year).
Drug: Cisplatin — Cisplatin 75* mg/m2 or 80* mg/m2, IV on Day 1 of each 21-day cycle up to 6 cycles.
  * 75 mg/m2 when in combination with pemetrexed, 80 mg/m2 when in combination with gemcitabine
Drug: Gemcitabine — Gemcitabine 1250 mg/m2, IV on Days 1 and 8 of each 21-day cycle up to 6 cycles
Drug: Pemetrexed — Pemetrexed 500 mg/m2, IV on Day 1 of each 21-day cycle up to 6 cycle

SUMMARY:
CP 751,871 is a fully human monoclonal antibody against the Insulin-Like Growth Factor 1 Receptor (IGF-1R). Preclinical and clinical data indicate that CP 751,871 augments the anti-tumor activity of chemotherapy. This study will identify the Maximal Tolerated Dose of CP 751,871 (or the Maximal Feasible Dose) in combination with standard gemcitabine-cisplatin chemotherapy for the treatment of advanced Non-Small Cell Lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven diagnosis of Stage IIIB (N3 and/or T4) or Stage IV Non-Small Cell Lung Cancer in patients 18-year-old or older, with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 not amenable to curative surgery or radiation therapy and an adequate organ function (bone marrow, hepatic, renal, and cardiac) within 14 days prior to enrollment.

Exclusion Criteria:

* Any prior treatment for Non-Small Cell Lung Cancer including chemotherapy, biologic response modifiers or therapy with any investigational agents.
* Patients with known brain metastases, spinal cord compression, uncontrolled superior vein cava syndrome or carcinomatous meningitis.
* Patients with gastrointestinal abnormalities including active gastrointestinal bleeding, pre-diabetes (pre-fasting glycemia > 120 g/dL and/or glycosylate haemoglobin level > 7.5%), known HIV or AIDS-related illness, significant active cardiac disease or receiving chronic steroid therapy or concurrent use of growth hormones or growth hormone inhibitors or aminoglycoside antibiotics should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Pfizer Investigational Site, Charleroi, Belgium
- Pfizer Investigational Site, Dublin, Ireland
- Spain (2):
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla

RESULTS

PARTICIPANT FLOW:
Groups:
- Figitumumab 6 mg/kg: Figitumumab 6 milligram (mg)/kilogram (kg) was administered intravenously (IV) on Day 1 of each cycle over 2.5 hours (hr) up to 6 cycles. Gemcitabine 1250 mg/meter square (m^2) was administered IV over approximately 30 minutes (min) on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 10 mg/kg: Figitumumab 10 mg/kg was administered IV on Day 1 of each cycle over 2.5 hr up to 6 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 20 mg/kg Dose Escalation: Figitumumab 20 mg/kg, was administered IV on Day 1 of each cycle over 2.5 hr up to 6 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 20 mg/kg RP2D Expansion 1.0 Infusion: The recommended phase 2 dose (R2PD) of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 1 hr up to 17 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 20 mg/kg RP2D Expansion 2.5 Infusion: The RP2D of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 2.5 hr up to 17 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 20 mg/kg Pemetrexed Expansion: The RP2D of figitumumab 20 mg/kg, was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 2.5 hr up to 17 cycles. Pemetrexed 500 mg/m^2 was administered IV over 10 min on Day 1 of each 21-day cycle up to 6 cycles. Cisplatin 75 mg/m^2 was administered IV over approximately 2 hr, following the completion of the pemetrexed treatment on Day 1 of each cycle up to 6 cycles.
Period: Overall Study
Arm/Group | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg Dose Escalation | Figitumumab 20 mg/kg RP2D Expansion 1.0 Infusion | Figitumumab 20 mg/kg RP2D Expansion 2.5 Infusion | Figitumumab 20 mg/kg Pemetrexed Expansion
Started | 6 | 3 | 6 | 10 | 8 | 13
Treated | 6 | 3 | 6 | 10 | 7 | 13
Completed | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 6 | 3 | 6 | 10 | 7 | 13
Not completed — Death | 4 | 1 | 4 | 5 | 1 | 10
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other | 2 | 2 | 2 | 3 | 3 | 3
Not completed — Enrolled, not treated | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants who received figitumumab 6, 10, 20 mg/kg and at the RP2D of 20 mg/kg with increasing infusion rates in combination with standard doses of gemcitabine and cisplatin. Participants who received figitumumab at the RP2D in combination with pemetrexed and cisplatin.
Arm/Group | All Participants
Number analyzed (Participants) | 45
Age Continuous [Mean (Standard Deviation); unit: Years] | 59.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT)
Description: Cycle 1 figitumumab attributed: Grade (Gr) 4 neutropenia (absolute neutrophil count <500 cells/cubic millimeter [mm^3]) >=7 days, febrile neutropenia (Gr 3, fever >=38.5 degrees Celsius), neutropenic infection (Gr 3 neutropenia, infection); Gr 4 thrombocytopenia (platelet <25,000 cells/mm^3), Gr 3 thrombocytopenia >=7 days/bleeding; other Gr 3 not blood/bone marrow Common Terminology Criteria for Adverse Events bar gastrointestinal toxicity, treatment-managed hyperglycemia/fatigue, hypersensitivity; Gr 3-4 hyperglycemia despite treatment; fail to adequately recover to continue study treatment
Time Frame: Start of treatment up to end of Cycle 1, Day 21
Population: Safety analysis set: All enrolled participants in the dose escalation who received at least 1 dose of study medication.
Measure: Number; unit: participants
Groups:
- Figitumumab 6 mg/kg: Figitumumab 6 mg/kg, was administered IV on Day 1 of each cycle over 2.5 hr up to 6 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 10 mg/kg: Figitumumab 10 mg/kg, was administered IV on Day 1 of each cycle over 2.5 hr up to 6 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 20 mg/kg Dose Escalation: Figitumumab 20 mg/kg was administered IV on Day 1 of each cycle over 2.5 hr up to 6 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
Arm/Group | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg Dose Escalation
Number analyzed (Participants) | 6 | 3 | 6
participants | 0 | 0 | 1

2. Secondary Outcome: Concentration at the End of Infusion (Cinf) for Figitumumab
Description: Figitumumab pharmacokinetic (PK) data was analyzed using noncompartmental methods
Time Frame: Cycle 1 for dose escalation and Cycle 4 for dose expansion
Population: PK analysis set: All enrolled participants who started treatment and had on-study samples to provide interpretable results.
Measure: Mean (Standard Deviation); unit: mg/liter (L)
Groups:
- Figitumumab 6 mg/kg: Figitumumab 6 mg/kg was administered IV on Day 1 of each cycle over 2.5 hr up to 6 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 20 mg/kg Expansion: The RP2D of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 2.5 to 1 hr up to 17 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
Arm/Group | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg Dose Escalation | Figitumumab 20 mg/kg Expansion
Number analyzed (Participants) | 5 | 1 | 4 | 13
mg/liter (L) | 120.4 (26.690) | 137.0 (NA) — Data available from only 1 participant | 435.0 (129.01) | 513.4 (136.58)

3. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Figitumumab
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). Figitumumab PK data was analyzed using noncompartmental methods
Time Frame: 0 (pre-dose), 1, 24, 72, 168, 336, 504 hr in Cycle 1 for dose escation and 0 (pre-dose), 1, 24, 72, 168, 336, 504 hr in Cycle 4 for expansion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg Dose Escalation | Figitumumab 20 mg/kg Expansion
Number analyzed (Participants) | 5 | 1 | 4 | 12
mg*hr/L | 26020 (6780.6) | 21500 (NA) — Data available from only 1 participant | 84100 (18983) | 121200 (50493)

4. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin) for Figitumumab
Description: Concentration at the end of Cycle 4
Time Frame: 0 (pre-dose) in Cycle 5 Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Figitumumab 20 mg/kg Expansion: The RP2D of figitumumab 20 mg/kg was administered IV on Day 1 of each cycle over 2.5 to 1 hr up to 17 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
Arm/Group | Figitumumab 20 mg/kg Expansion
Number analyzed (Participants) | 11
mg/L | 113.6 (47.266)

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Cisplatin
Description: Cisplatin PK data was analyzed using noncompartmental methods. Plasma exposure parameters for cisplatin were analyzed in the absence (Cycle 1) and presence of (Cycle 2) figitumumab
Time Frame: 0 (pre-dose), 1.917, 2.5, 3, 4, 5, 24 hr on Cycle 1, Day 1 and Cycle 2, Day 1 for cisplatin 75 mg/m^2 and 0 (pre-dose), 0.917, 1.5, 2, 3, 4, 23 hr on Cycle 1, Day 1 and Cycle 2, Day 1 for cisplatin 80 mg/m^2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram (ng)/mL
Groups:
- Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 1); Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 2): The RP2D of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 2.5 to 1 hr up to 17 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 1); Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 2): The RP2D of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 2.5 hr up to 17 cycles. Pemetrexed 500 mg/m^2 was administered IV over 10 min on Day 1 of each 21-day cycle up to 6 cycles. Cisplatin 75 mg/m^2 was administered IV over approximately 2 hr, following the completion of the pemetrexed treatment on Day 1 of each cycle up to 6 cycles.
Arm/Group | Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 1) | Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 2) | Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 1) | Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 2)
Number analyzed (Participants) | 15 | 11 | 13 | 11
nanogram (ng)/mL | 3.816 (1.5485) | 3.880 (0.8490) | 2.845 (0.8804) | 3.490 (1.1435)

6. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Cisplatin
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). Cisplatin PK data was analyzed using noncompartmental methods. Plasma exposure parameters for cisplatin were analyzed in the absence (Cycle 1) and presence (Cycle 2) of figitumumab
Time Frame: as for outcome 5
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/L
Arm/Group | Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 1) | Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 2) | Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 1) | Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 2)
Number analyzed (Participants) | 15 | 11 | 13 | 11
ng*hr/L | 38.23 (7.2762) | 45.18 (15.005) | 37.12 (8.7975) | 48.29 (13.931)

7. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Gemcitabine
Description: Gemcitabine PK data was analyzed using noncompartmental methods. Plasma exposure parameters for gemcitabine were analyzed in the absence (Cycle) 1 and presence (Cycle 2) of figitumumab
Time Frame: 0 (pre-dose), 0.417, 1, 1.5, 2.5, 3.5 hr on Cycle 1, Day 1 and Cycle 2, Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/L
Groups:
- Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 2): The RP2D of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 (absence) and on Day 1 of each cycle (presence) thereafter over 2.5 to 1 hr up to 17 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
Arm/Group | Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 1) | Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 2)
Number analyzed (Participants) | 15 | 9
ng/L | 12.85 (6.9644) | 23.97 (18.764)

8. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Gemcitabine
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). Gemcitabine PK data was analyzed using noncompartmental methods. Plasma exposure parameters for gemcitabine were analyzed in the absence (Cycle 1) and presence (Cycle 2) of figitumumab
Time Frame: 0 (pre-dose), 0.417, 1, 1.5, 2.5, 3.5 hr on Cycle 1, Day 1 and Cycle 2, Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/L
Arm/Group | Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 1) | Cisplatin 80 mg/m^2/Gemcitabine Expansion (Cycle 2)
Number analyzed (Participants) | 15 | 9
ng*hr/L | 6.665 (3.0299) | 12.53 (7.5062)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Pemetrexed
Description: Pemetrexed PK data was analyzed using noncompartmental methods. Plasma exposure parameters for pemetrexed were analyzed in the absence (Cycle 1) and presence (Cycle 2) of figitumumab
Time Frame: 0, 0.167, 1.167, 2.167, 4.167, 6.167, 24.167 hr on Cycle 1, Day 1 and Cycle 2, Day 1 for pemetrexed 500 mg/m^2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 1) | Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 2)
Number analyzed (Participants) | 13 | 11
ng/mL | 72.96 (25.581) | 93.13 (12.560)

10. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Pemetrexed
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast). Pemetrexed PK data was analyzed using noncompartmental methods. Plasma exposure parameters for pemetrexed were analyzed in the absence (Cycle 1) and presence (Cycle 2) of figitumumab
Time Frame: 0, 0.167, 1.167, 2.167, 4.167, 6.167, 24.167 hr on Cycle 1, Day 1 and Cycle 2, Day 1 for pemetrexed 500 mg/m^2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*hr/L
Arm/Group | Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 1) | Cisplatin 75 mg/m^2/Pemetrexed Expansion (Cycle 2)
Number analyzed (Participants) | 13 | 11
ng*hr/L | 132.2 (71.512) | 161.6 (39.335)

11. Secondary Outcome: Percentage of Participants With Objective Response or Prolonged Stabilization
Description: Percentage of participants with a confirmed complete response (CR), confirmed partial response (PR), or stable disease (SD) for at least 12 weeks on study according to Response Evaluation Criteria in Solid Tumors (RECIST). Participants with non measurable disease were considered having a clinical benefit response only in the case of achievement of CR. Participants who developed early progressive disease post dosing and prior to response evaluation were considered to have progressed on study. Confirmed responses were those that persisted on repeat imaging >= 4 weeks after initial response
Time Frame: Screening, from Cycle 2 onwards computerized tomography (CT) scan done within 7-10 days prior to next cycle (approximately Day 15 of each cycle), follow-up (30 days after last study treatment dose)
Population: Efficacy analysis set: All participants with measurable disease at baseline, receiving at lesast 1 dose of figitumumab with a response assessment made by the investigator according to the RECIST system.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Overall Population: Participants who received figitumumab 6, 10, 20 mg/kg and at the RP2D of 20 mg/kg with increasing infusion rates in combination with standard doses of gemcitabine and cisplatin. Participants who received figitumumab at the RP2D in combination with pemetrexed and cisplatin.
- Figitumumab 20 mg/kg With Gemcitabine and Cisplatin: The RP2D of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 2.5 to 1 hr up to 17 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 20 mg/kg Expansion With Pemetrexed: The RP2D of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 2.5 hr up to 17 cycles. Pemetrexed 500 mg/m^2 was administered IV over 10 min on Day 1 of each 21-day cycle up to 6 cycles. Cisplatin 75 mg/m^2 was administered IV over approximately 2 hr, following the completion of the pemetrexed treatment on Day 1 of each cycle up to 6 cycles.
Arm/Group | Overall Population | Figitumumab 20 mg/kg With Gemcitabine and Cisplatin | Figitumumab 20 mg/kg Expansion With Pemetrexed
Number analyzed (Participants) | 45 | 23 | 13
Percentage of participants | 53.3 [37.9 to 68.3] | 56.5 [34.5 to 76.8] | 46.2 [19.2 to 74.9]

12. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time from the date of enrollment to date of documented disease progression, or death due to any cause
Time Frame: Screening, from Cycle 2 onwards CT scan done within 7-10 days prior to next cycle (approximately Day 15 of each cycle), follow-up (30 days after last study treatment dose)
Population: as for outcome 11
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Overall Population | Figitumumab 20 mg/kg With Gemcitabine and Cisplatin | Figitumumab 20 mg/kg Expansion With Pemetrexed
Number analyzed (Participants) | 40 | 21 | 10
months | 5.7 [2.0 to 6.5] | 6.5 [1.7 to 10.2] | 5.4 [1.6 to 5.7]

13. Secondary Outcome: Duration of Response (DR)
Description: For responding patients (CR and PR): Time from the date that CR or PR was first recorded to the date of the first documentation of progression
Time Frame: as for outcome 12
Population: No analysis of this parameter was performed. Due to the exploratory nature of the study, the analysis of the efficacy of figitumumab was limited to the assessment of clinical benefit response and PFS.
Groups:
- Overall Population With PR and CR: Participants with PR and CR who received figitumumab 6, 10, 20 mg/kg and at the RP2D of 20 mg/kg with increasing infusion rates in combination with standard doses of gemcitabine and cisplatin. Participants with PR and CR who received figitumumab at the RP2D in combination with pemetrexed and cisplatin.
Arm/Group | Overall Population With PR and CR
Number analyzed (Participants) | 0

14. Secondary Outcome: Percentage of Participants With Blood Anti-drug Antibody (ADA) Specific for Figitumumab
Description: Percentage of participants with positive total or neutralizing anti-drug antibody (ADA) for figitumumab
Time Frame: 30 min prior to figitumumab infusion in Cycle 1 and Cycle 4, end of study, fourth follow up visit (approximately 150 days after last dose)
Population: ADA analysis set: All enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Groups:
- Figitumumab 20 mg/kg RP2D Expansion 1.0 Infusion: The RP2D of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 1 hr up to 17 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 20 mg/kg RP2D Expansion 2.5 Infusion: The RP2D of igitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 2.5 hr up to 17 cycles. Gemcitabine 1250 mg/m^2 was administered IV over approximately 30 min on Day 1 and Day 8 of each 21-day cycle up to 6 cycles. Cisplatin 80 mg/m^2 was administered IV over approximately 1 hr, following the completion of the gemcitabine treatment on Day 1 of each cycle up to 6 cycles.
- Figitumumab 20 mg/kg Pemetrexed Expansion: The RP2D of figitumumab 20 mg/kg was administered IV 24 hr after start of cisplatin infusion in Cycle 1 and on Day 1 of each cycle thereafter over 2.5 hr up to 17 cycles. Pemetrexed 500 mg/m^2 was administered IV over 10 min on Day 1 of each 21-day cycle up to 6 cycles. Cisplatin 75 mg/m^2 was administered IV over approximately 2 hr, following the completion of the pemetrexed treatment on Day 1 of each cycle up to 6 cycles.
Arm/Group | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg Dose Escalation | Figitumumab 20 mg/kg RP2D Expansion 1.0 Infusion | Figitumumab 20 mg/kg RP2D Expansion 2.5 Infusion | Figitumumab 20 mg/kg Pemetrexed Expansion
Number analyzed (Participants) | 6 | 3 | 6 | 10 | 7 | 13
Percentage of participants
  C1D1 - Negative | 50.0 | 33.3 | 50.0 | 80.0 | 100 | 100
  C1D1 - Positive | 0 | 0 | 0 | 0 | 0 | 0
  C1D1 - Not determined | 50.0 | 66.7 | 50.0 | 20.0 | 0 | 0
  C4D1 - Negative | 16.7 | 0 | 50.0 | 30.0 | 71.4 | 53.8
  C4D1 - Positive | 0 | 0 | 0 | 0 | 0 | 0
  C4D1 - Not determined | 83.3 | 100 | 50.0 | 70.0 | 28.6 | 46.2
  End of Study - Negative | 83.3 | 0 | 50.0 | 20.0 | 42.9 | 46.2
  End of Study - Positive | 0 | 0 | 0 | 0 | 0 | 0
  End of Study - Not determined | 16.7 | 100 | 50.0 | 80.0 | 51.7 | 53.8
  Follow Up - Negative | 0 | 0 | 0 | 0 | 14.3 | 0
  Follow Up - Positive | 0 | 0 | 0 | 0 | 0 | 0
  Follow Up - Not determined | 100 | 100 | 100 | 100 | 85.7 | 100

15. Secondary Outcome: Serum Total Circulating Insulin-like Growth Factor (IGF-1) Levels
Description: To monitor serum total IGF-1 levels as a potential pharmacodynamic response to figitumumab treatment
Time Frame: Baseline, Day 8, end of study
Population: Biomarker analysis set: All enrolled participants who received at least 1 dose of study medication.
Measure: Mean (Inter-Quartile Range); unit: ng/mL
Arm/Group | Overall Population
Number analyzed (Participants) | 40
ng/mL
  Baseline | 124.88 [91 to 143]
  End of study | 543.63 [343 to 694]

16. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD)
Description: The MTD was defined as the highest dose level below the maximum administered dose which caused 0 or 1 out of 6 participants to experience a DLT in that given cohort at Cycle 1
Time Frame: Cycle 1, up to Day 21
Population: Safety analysis set: All enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: mg/kg
Arm/Group | Overall Population
Number analyzed (Participants) | 45
mg/kg | 20

17. Other Pre Specified Outcome: Recommended Phase 2 Dose (RP2D)
Description: The RP2D was determined after review and discussion by sponsor and investigators of the study data. Consideration was given to type and severity of toxicity as well as clinical suitability for long-term administration
Time Frame: Baseline to end of dose escalation, which was assessed in the last participant of the dose escalation portion of the study in Month 19
Population: Safety analysis set: All enrolled participants who received at least 1 dose of study medication.
Measure: Number; unit: mg/kg
Groups:
- Overall Participapnts: Participants who received figitumumab 6, 10, 20 mg/kg and at the RP2D of 20 mg/kg with increasing infusion rates in combination with standard doses of gemcitabine and cisplatin. Participants who received figitumumab at the RP2D in combination with pemetrexed and cisplatin.
Arm/Group | Overall Participapnts
Number analyzed (Participants) | 45
mg/kg | 20

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (AE) were reported from the time of the first dose of study treatment up to 150 days after the last dose of study treatment.
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Figitumumab 6 mg/kg | Figitumumab 10 mg/kg | Figitumumab 20 mg/kg Dose Escalation | Figitumumab 20 mg/kg RP2D Expansion 1.0 Infusion | Figitumumab 20 mg/kg RP2D Expansion 2.5 Infusion | Figitumumab 20 mg/kg Pemetrexed Expansion
Serious Adverse Events (participants affected / at risk) | 3/6 | 2/3 | 3/6 | 7/10 | 2/7 | 8/13
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 6/6 | 10/10 | 7/7 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 6 mg/kg (N=6) | Figitumumab 10 mg/kg (N=3) | Figitumumab 20 mg/kg Dose Escalation (N=6) | Figitumumab 20 mg/kg RP2D Expansion 1.0 Infusion (N=10) | Figitumumab 20 mg/kg RP2D Expansion 2.5 Infusion (N=7) | Figitumumab 20 mg/kg Pemetrexed Expansion (N=13)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 1 | 2
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Carbon dioxide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arterial thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Figitumumab 6 mg/kg (N=6) | Figitumumab 10 mg/kg (N=3) | Figitumumab 20 mg/kg Dose Escalation (N=6) | Figitumumab 20 mg/kg RP2D Expansion 1.0 Infusion (N=10) | Figitumumab 20 mg/kg RP2D Expansion 2.5 Infusion (N=7) | Figitumumab 20 mg/kg Pemetrexed Expansion (N=13)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 3 | 2 | 5 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 1 | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 5 | 3 | 5 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1 | 2 | 2 | 3 | 5
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 2
Motion sickness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ototoxicity (Ear and labyrinth disorders) | 1 | 0 | 3 | 3 | 2 | 3
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 2 | 1 | 1 | 2
Conjunctivitis (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 3
Keratoconjunctivitis sicca (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 3 | 2 | 4 | 3
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 3 | 3 | 1 | 6
Diverticular perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Lip haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 1 | 4 | 5 | 5 | 8
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 4 | 2 | 4 | 5
Asthenia (General disorders) | 4 | 2 | 5 | 6 | 5 | 6
Chest pain (General disorders) | 3 | 0 | 2 | 2 | 1 | 4
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 2 | 2 | 2 | 1 | 0 | 4
Fatigue (General disorders) | 3 | 1 | 2 | 2 | 4 | 4
Hypothermia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 3 | 1 | 2 | 5 | 3 | 3
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Performance status decreased (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 3 | 3 | 3 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 2
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time shortened (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 3 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 0 | 1
Blood albumin decreased (Investigations) | 0 | 0 | 1 | 3 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Blood chloride decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 3 | 0 | 1 | 3 | 3 | 6
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood immunoglobulin A decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood immunoglobulin G decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 1 | 1 | 1 | 0 | 0
Blood magnesium increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 1 | 0 | 1 | 2 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 1 | 1 | 1 | 3
Glucose urine present (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Glutamate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 1 | 1 | 2 | 0 | 2
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
Platelet count decreased (Investigations) | 3 | 1 | 2 | 2 | 2 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 2 | 1 | 1
White blood cell count decreased (Investigations) | 2 | 1 | 1 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0 | 5 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2 | 5 | 5 | 4 | 10
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 2
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 3 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 3 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 2 | 0 | 1 | 0 | 2 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1
Hypokinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0 | 3 | 2 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0 | 1 | 2
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 3 | 2 | 5
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2 | 1 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 3 | 0 | 2
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 2
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 1 | 0 | 2 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
A total of 46 patients were enrolled in this study but only 45 of them were evaluable because 1 patient was enrolled but did not participate due to early symptomatic deterioration prior to starting treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.